CLINICAL TRIAL: NCT07182630
Title: Investigation Of The Effects Of Anti-Tnf-Α And Non-Tnf-Α Drugs On Aerobic Capacity, Muscle Strength, Fatigue, Cardiovascular Disease Risk Factors, And Disease Activity İn Patients With Rheumatoid Arthritis
Brief Title: Investigation Of The Effects Of Anti-Tnf-Α And Non-Tnf-Α Drugs İn Patients With Rheumatoid Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Ahmet Seçkin Korkmaz, Principal Investigator, Firat University
Other Study IDs: FU-FTR-ASK-01
Record Dates: First submitted 2025-08-18; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Rheumatoid Arthritis (RA
Keywords: Anti TNF-α; Non TNF-α; Rheumatoid arthritis; Aerobic Capacity
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People Using Anti-TNF-α Medication: 20 participants will consist of patients using anti-TNF-α drugs.
- People Using Non-TNF-α Medication: 20 participants will consist of patients using non-TNF-α drugs.

SUMMARY:
In RA, joint structure is damaged due to destructive inflammation in the synovium. This condition negatively affects the patient's level of physical activity. As the patient becomes more immobile, their muscle mass and strength decrease and their aerobic capacity declines. One of the drug groups used in the pharmacological treatment of RA is anti-TNF-α drugs. The aim of this study is to investigate the effects of anti-TNF-α and non-TNF-α drug treatments on aerobic capacity, muscle strength, fatigue, cardiorespiratory risk factors, and disease activity in RA patients.

DETAILED DESCRIPTION:
The basic principle in the treatment of rheumatoid arthritis is to prolong the period of remission in patients. Even if complete remission is not achieved, improvements in symptoms and clinical findings enable patients to maintain their functional capacity at a certain level, which is important for their quality of life. To this end, a multidisciplinary approach involving exercise therapy, pharmacological treatment, and psychological support is applied. The primary goal of pharmacological treatment is to intervene in inflammatory pathways. While there are studies in the literature on the relationship of these pharmacological agents with other disease-related mediators and the clinical course of the disease, no studies have been found that examine the relationship between aerobic capacity, which is one of the basic indicators of the patient's functional level, and fatigue, cardiorespiratory risk factors, and quality of life, which are related to aerobic capacity. Based on the results of the study, the aim was to compare the effects of anti-TNF-α and non-TNF-α drugs on aerobic capacity, fatigue, muscle strength, cardiovascular disease risk factors, and disease activity in RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA according to the 2010 American College of Rheumatology (ACR-2010) criteria
* Be between 18 and 65 years of age
* Be literate
* Have been using one of the anti-TNF-α or non-TNF-α drugs for a period of 1-3 years

Exclusion Criteria:

* Being pregnant or having a diagnosis of malignancy
* Having a dysfunction that would limit physical activity (cycling for aerobic capacity assessment), such as severe neurological involvement, immobility, or incooperation
* Having a regular exercise habit (reporting a habit of exercising 3 or more days per week)
* Having another chronic disease
* Having cardiac symptoms according to the New York Heart Association
* Having mental problems that prevent participation in assessments

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants will be included in the study.
Study Population: The study will include 40 patients aged 18-65 who are being followed up at the Department of Rheumatology at Fırat University Hospital and who have been diagnosed with RA according to the 2010 RA criteria of the American College of Rheumatology (ACR).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximal Oxygen Consumption | First Day 1
  VO2max will be assessed using Cosmed FitMate Pro® (Cosmed, Italy). The FitMate Pro® includes a turbine flow meter to measure ventilation and a galvanic fuel cell oxygen sensor to analyze the oxygen fraction in exhaled gases. The FitMate Pro® performs self-calibration before each measurement. A face mask will be placed over the participant's face to sample exhaled air, which will then be connected to the turbine flow meter. After resting for 5 minutes (while seated on the ergometer), participants will be asked to begin pedaling on the bicycle ergometer (E200 Cosmed®, Italy) starting at 25W. The load will be increased by 25W every 3 minutes until exhaustion.

OTHER OUTCOMES:
Fatigue Severity Scale | First Day 1
  There are nine questions related to fatigue on this scale. Patients are asked to rate these questions on a scale of 1 to 7. The assessment results in a score between 9 and 63. A higher score indicates greater fatigue.
Sarcopenia assessment | First Day 1
  In the assessment of sarcopenia, patients' gross grip strength will be evaluated. Gross grip strength will be assessed using the Jamar Hand Dynamometer. The Jamar Hand Dynamometer is a method recommended by the American Association of Occupational Therapists (AAOT) for measuring hand grip strength, and is considered the gold standard with proven validity and reliability.
Cardiovascular Disease Risk Factors | First Day 1
  Cardiovascular risk factors will be assessed using Framingham risk factors. The risk factors assessed in the Framingham Risk Score are age, gender, total cholesterol level, HDL cholesterol level, systolic blood pressure/use of medication for high blood pressure, and smoking. In the Framingham Risk Score, patients are categorized into three groups: high, moderate, and low risk. Patients with a 10-year risk of adverse events >20% are considered high risk, those with a risk of 10-20% are considered moderate risk, and those with a risk of <10% are considered low risk.
Quality of Life Assessment | First Day 1
  The scale was developed for use in individuals with RA and is designed to be completed by the patients themselves. The scale consists of 30 questions, which are scored as "yes-1" and "no-0." The resulting scores range from 0 to 30, with higher scores indicating poorer quality of life.
Disease Activity Assessment | First Day 1
  The Disease Activity Score-28 (DAS-28) will be used to assess disease activity. Twenty-eight joints, including fingers, wrists, elbows, shoulders, and knees, are examined for tenderness and swelling. Patients are asked to assign a score between 0 and 100 for their overall well-being. Erythrocyte sedimentation rate (ESR) and C-reactive protein are determined, and DAS-28 is calculated using all of these data. High scores indicate high disease activity

CONTACTS AND LOCATIONS:
Overall Officials: Songül BAĞLAN YENTÜR, Doç. Dr., Study Director — Firat University
Locations (1):
- Fırat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No